CLINICAL TRIAL: NCT04388878
Title: A PHASE 1, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, STUDY TO ASSESS SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE AND MULTIPLE ASCENDING ORAL DOSES OF PF-07054894 IN HEALTHY ADULT PARTICIPANTS
Brief Title: Study Of Single And Multiple Ascending Doses Of PF-07054894 In Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: C4151001; 2020-000772-38 (EudraCT Number)
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PF-07054894 (Experimental): Participants will receive single or multiple ascending doses of oral PF-07054894
  Interventions: Drug: PF-07054894
- Placebo (Placebo Comparator): Participants will receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07054894 — Participants will receive oral ascending doses
  Arms: PF-07054894
Drug: Placebo — Participants will receive matching placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the safety, tolerability, and PK of single escalating doses and multiple escalating doses of PF-07054894.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (of non-child bearing potential) participants must be 18 to 55 years of age, inclusive, and with BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Male and female of non-child bearing potential participants who are overtly healthy as determined by medical evaluation.
* Participants must be willing to avoid direct sunlight exposure or any high intensity ultraviolet light exposure, from admission to FU1 and to apply sun screen/lotion with a high sun protection factor, as appropriate.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, immunological/rheumatological, or allergic diseases.
* Evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB), history of HIV infection, hepatitis B, or hepatitis C.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Have a history of systemic infection requiring hospitalization, parenteral antimicrobial therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 1.
* History of phototoxicity and photosensitivity.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
AEs following Single ascending dose (SAD) | Day 1 up to Day 28 (SAD)
  Frequency, severity and causal relationship of treatment emergent adverse events (TEAEs) and withdrawals due to TEAEs
AEs following multiple ascending dose (MAD) | Day 1 up to Day 42 (MAD)
  Frequency, severity and causal relationship of treatment emergent adverse events (TEAEs) and withdrawals due to TEAEs
Percentage of subjects with laboratory abnormalities | Day 1 up to Day 7 (SAD) or Day 1 up to Day 21 (MAD)
Number of subjects with change from baseline in vital signs | Day 1 up to Day 7 (SAD) or Day 1 up to Day 21 (MAD)
  Number of subjects with change from baseline of blood pressure, pulse rate, and oral temperature
Number of subjects with change from baseline in electrocardiogram (ECG) parameters | Day 1 up to Day 7 (SAD) or Day 1 up to Day 21 (MAD)

SECONDARY OUTCOMES:
Maximum Plasma concentration (Cmax) | Day 1 (SAD) or Day 1 and Day 14 (MAD)
  Maximum observed plasma concentration (Cmax)
Time to reach plasma Cmax (Tmax) | Day 1 (SAD) or Day 1 and Day 14 (MAD)
  Time to reach maximum observed plasma concentration (Tmax)
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Day 1 up to Day 3 (SAD)
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] | Day 1 up to Day 3 (SAD)
  AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞).
Dose normalized Cmax (Cmax(dn)) | Day 1 (SAD) or Day 1 and Day 14 (MAD)
  Dose normalized maximum plasma concentration (Cmax(dn))
Apparent Oral Clearance (CL/F) | Day 1 (SAD) or Day 14 (MAD)
  Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed and a quantitative measure of the rate at which the drug is removed from the blood.
Apparent Volume of Distribution (Vz/F) | Day 1 (SAD) or Day 14 (MAD)
  Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Single dose and Multiple Dose PK half-life (t½) | Day 1 (SAD) or Day 14 (MAD)
  Plasma elimination half-life is the time measured for the plasma concentration to decrease by one half.
Observed Accumulation Ratio for Cmax (Rac,Cmax) | MAD, Day 14
  Accumulation ratio based on maximum plasma concentration (Cmax) calculated as: Rac,Cmax = Cmax at steady state (ss) divided by Cmax at first dose.
Observed Accumulation Ratio for AUCτau (Rac, AUCτau) | MAD, Day 14
  Accumulation ratio calculated as, Rac obtained from Area Under the Concentration Time Curve (AUCτau) from time 0-τau (Day 14) divided by AUC from time 0-τau (Day 1).
Area Under the Curve From Time Zero to End of Dosing Interval (AUCτau) | Day 1 and Day 14 of MAD
  Area under the concentration curve from time 0 to end of dosing interval (AUCτau), where dosing interval is 12 hours.
Minimum Observed Plasma Trough Concentration (Cmin) | Day 1 up to Day 14 of MAD
  Minimum plasma concentration over the dosing interval τau (12 hour) from first dose to last dose
Multiple dose PK/AUCτau (dn) | Day 1 and Day 14 of MAD
  Dose normalized area under the curve over the dosing interval τau (12 hour) after the first and last dose (AUCτau (dn))
Cumulative Amount of Drug Recovered Unchanged in Urine during dosing interval (Ae,τau) | MAD, Day 14
  Cumulative amount of drug recovered unchanged in urine during the dosing interval, where the dosing interval is 12 hours (Ae,τau)
Percentage of Dose Recovered Unchanged in Urine From Time 0 to the Dosing Interval τau (Ae,τau%) | MAD, Day 14
  Percent of dose recovered in urine as unchanged drug over the dosing interval (Ae,τau%)
Renal Clearance (Clr) | MAD, Day 14
  Renal clearance calculated as cumulative amount of drug recovered unchanged in urine during the dosing interval (Ae,τau) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCτau), where dosing interval is 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4151001